CLINICAL TRIAL: NCT02340468
Title: Breast Tumor Oxygenation During Exercise
Status: Withdrawn | Type: Observational
Why Stopped: Not clinical trial
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg,Ph.D.,Director, Beckman Laser Institute and Medical Clinic and Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 20141505
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: diffuse optical spectroscopy — diffuse optical spectroscopy

SUMMARY:
In the field of cancer treatment, it is generally accepted that the enhancement of oxygen delivery to tumors can augment the effect of anti-cancer therapies. In the case of chemotherapy, this enhancement might lead to a larger amount of a given dose of treatment reaching the tumor and having an effect.

DETAILED DESCRIPTION:
While the benefits of exercise on overall health are widely documented, little is known about how exercise affects the progression or treatment of malignant neoplasms. Tumors have a complex vascular network which is likely affected by the global changes in hemodynamics and perfusion that occur during moderate exercise. Increased tumor oxygenation is clinically relevant as it may counteract the hypoxic tumor environment which is known to contribute to resistance to chemo- and radiation therapies, angiogenesis, invasiveness and metastasis, genomic instability, and resistance to cell death.

The researcher can use noninvasive optical imaging technology called diffuse optical spectroscopy to safely and non-invasively quantify the dynamics of blood flow and metabolism in tumors and normal tissue of subjects undergoing supervised cycling exercise. The researcher can determine that exercise will measurably increase tumor oxygenation, and that this effect will be proportional to the intensity and/or duration of the exercise performed.

ELIGIBILITY:
Inclusion Criteria:

* Tumor group, female, Greater than 21 years of age but less than 70 years of age, Current diagnosis of breast cancer stage 0 - IV or radiologically suspicious for breast cancer BI-RADS score 4 or 5.
* Control group,Female, Greater than 21 years of age but less than 70 years of age, Not currently diagnosed with breast cancer

Exclusion Criteria:

* Under 21 years of age, Pregnant or breastfeeding, Contraindications for moderate exercise, history of heart, pulmonary, or musculoskeletal disease; physician instructions to restrict physical activity.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be recruited from an outpatient at UC Irvine Health
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Measure breast tumor oxygenation | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tromberg, PhD, Principal Investigator — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute Medical Clinic, Irvine, California, United States